CLINICAL TRIAL: NCT05628415
Title: Comparison Between the Non-powered AEON™ Endostapler and Echelon FLEX™ Powered Plus Stapler With Regards to the Closure of Lung Tissue After Lung Resection in the Presence of Severe Lung Emphysema: A Prospective Randomized Single-blinded Monocentric Study
Brief Title: Comparison Between the Non-powered AEON™ Endostapler and Echelon FLEX™ Powered Plus Stapler With Regards to the Closure of Lung Tissue After Lung Resection in the Presence of Severe Lung Emphysema
Acronym: Stapler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-D0079; kt22Lardinois3
Record Dates: First submitted 2022-11-15; First posted 2022-11-28 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Air Leak; Lung Resection
Keywords: severe lung emphysema; AEON™ Endostapler; Echelon FLEX™ Powered plus Stapler; lung-volume-reduction-surgery (LVRS)
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Intervention Model Description: prospective randomized single-blinded monocentric study
Who Masked: Participant
Masking Description: Only the Patient is blinded to the study. Patients do not know which stapler they are being treated with on which side because they are under anesthesia in the operating room and also do not have access to information regarding the stapler being used afterwards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procedure: non-powered AEON™ Endostapler (Active Comparator): Bilateral or unilateral lung-volume-reduction-surgery (LVRS) by video-assisted thoracic surgery (VATS) or open method with use of the non-powered AEON™ Endostapler for left and/or right side of the lung. By randomization it is specified on which side and with which method the lung tissue will be closed. If bilateral surgery is planned, the other side is automatically closured using the other method. In cases of a unilateral surgery a random stapler as stated in the envelop would be allocated for that side in question.
  Interventions: Procedure: Non-powered AeonTM Endostapler (according to manufacturer medical device classification IIb)
- Procedure: Echelon FLEX™ Powered plus Stapler (Active Comparator): Bilateral or unilateral lung-volume-reduction-surgery (LVRS) by video-assisted thoracic surgery (VATS) or open method with use of the Echelon FLEX™ Powered plus Stapler for left and/or right side of the lung. By randomization it is specified on which side and with which method the lung tissue will be closed. If bilateral surgery is planned, the other side is automatically closured using the other method. In cases of a unilateral surgery a random stapler as stated in the envelop would be allocated for that side in question.
  Interventions: Procedure: Echelon FLEX™ Powered plus Stapler (according to manufacturer medical device classification IIb)

INTERVENTIONS:
Procedure: Non-powered AeonTM Endostapler (according to manufacturer medical device classification IIb) — Closure of the left and/or right side of the lung after bilateral or unilateral lung-volume-reduction- surgery is performed with the non-powered Aeon™ Endostapler (Lexington medical) 60-mm and 45-mm. At the end of the operation, two 24F apical chest tubes are placed on each side and are systematically set at -10 cm H2O suction via the Medela- Topaz™ system. Air leak will be measured quantitatively in ml per minute by use of a Medela-Topaz™ system. Cessation of air leak is the case when a value of 0ml/min or two consecutive values under 30 ml/min by use of thoracic drainage Medela- Topaz™ system are read.
  Arms: Procedure: non-powered AEON™ Endostapler
Procedure: Echelon FLEX™ Powered plus Stapler (according to manufacturer medical device classification IIb) — Closure of the left and/or right side of the lung after bilateral or unilateral lung-volume-reduction- surgery is performed with the Echelon FLEX™ Powered plus Stapler (Ethicon) 60-mm and 45-mm. At the end of the operation, two 24F apical chest tubes are placed on each side and are systematically set at -10 cm H2O suction via the Medela- Topaz™ system. Air leak will be measured quantitatively in ml per minute by use of a Medela-Topaz™ system. Cessation of air leak is the case when a value of 0ml/min or two consecutive values under 30 ml/min by use of thoracic drainage Medela- Topaz™ system are read.
  Arms: Procedure: Echelon FLEX™ Powered plus Stapler

SUMMARY:
Prolonged air leak is reported in up to 60 to 75% of patients after lung operation in the presence of severe lung emphysema. The effect of the non-powered AEONTM Endostapler as compared to the Echelon FlexTM Powered plus stapler on the volume and duration of air leak and on the time to chest drain removal after lung operation in the presence of severe lung emphysema will be investigated in a randomized, prospective, single-blinded clinical trial.

DETAILED DESCRIPTION:
Patients with severe lung emphysema Grad III or IV scheduled for an operation by video-assisted thoracic surgery (VATS) or open method at the Department of Thoracic Surgery at the University Hospital Basel will be pre-screened in terms of inclusion and exclusion criteria. Before the operation, a randomization envelope is opened in the operation room, in which it is specified on which side and with which method the lung tissue will be closed. If bilateral surgery is planned, the other side is automatically closured using the other method. If for example the non-powered AEONTM Endostapler is randomly allocated to the left side, the right side is automatically operated with the Echelon FLEXTM Powered plus Stapler and vice versa. In cases of a unilateral surgery a random stapler as stated in the envelop would be allocated for that side in question. On the day of the operation, postoperative air leak will be measured quantitatively in ml per minute immediately, 2h, 4h, 8h, and 12h after skin closure. Starting on the first postoperative day, this is done twice a day at 8 am and 5 pm until the air leak stops or another surgery must be performed. Cessation of air leak is the case when a value of 0ml/min or two consecutive values under 30 ml/min by use of thoracic drainage Medela- Topaz™ system are read by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Patients discussed in the interdisciplinary emphysema treatment board and found to have the indication for a LVRS or patients who meet the criteria in agreement with pneumology recommendation for bilateral or unilateral LVRS with pulmonary emphysema (all morphologies including chronic obstructive pulmonary disease (COPD) GOLD III and IV) or patients operated for other Pathology other than lung emphysema requiring lung resection in the presence of severe lung emphysema.

Exclusion Criteria:

* non-bullous pulmonary emphysema
* Severely impaired carbon monoxide diffusing capacity (≤ 20% of predicted value, One-second capacity (FEV1) ≤ 20% of predicted value with a homogeneous emphysema morphology
* Patients with severe pulmonary arterial hypertension (mPAP > 35 mmHg) and are symptomatic
* Significant (i.e. clinically relevant and symptomatic) Coronary Arterial Disease (CAD)
* Inability to follow the procedures of the study, e. g. due to language problems, psychological disorders, dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent person
* Current enrolment in another clinical trial studying an experimental treatment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Time interval between the end of operation (skin closure) and air leak closure (when the volume is < 30 ml/min measured twice on Medela- Topaz™ drainage system) between the two staplers. | End of the operation (0 hours) until timepoint of air leak closure (approx. 3 days to a maximum of 7 days)
  Comparison of the time interval between the end of operation (skin closure) and air leak closure (when the volume is < 30 ml/min measured twice on drainage system) between the two staplers.
Change in Volume of air leak | End of the operation (0 hours), at 2 hours, 4 hours, 8 hours and 12 hours thereafter and from the first postoperative day, at 8 am and 5 pm daily until removal of the chest tubes (approx. 3 days to a maximum of 7 days)
  Volume of air leak measured following connection of chest tube drainages until removal of the chest tubes

SECONDARY OUTCOMES:
Number of postoperative air leaks | End of the operation (0 hours) until timepoint of air leak closure (approx. 3 days to a maximum of 7 days)
  Number of postoperative air leaks
Duration of postoperative air leaks until removal of the chest tubes in days | End of the operation (0 hours) until timepoint of air leak closure (approx. 3 days to a maximum of 7 days)
  Duration of postoperative air leaks until removal of the chest tubes in days
Postoperative complications graded using the Clavien -Dindo Classification | End of the operation (0 hours) until timepoint of air leak closure (approx. 3 days to a maximum of 7 days)
  The Clavien Classification system differentiates in five degrees of severity upon the intention to treat (Grade-I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions up to Grade-V: Death of a patient).
Number of resurgeries due to prolonged or profuse air leak | From the day of admittance to hospital to the day of discharge (approx. 7 days)
  Number of resurgeries due to prolonged or profuse air leak

CONTACTS AND LOCATIONS:
Overall Officials: Didier Lardinois, Prof. Dr. med., Study Director — Department of Thoracic Surgery, University Hospital Basel
Locations (1):
- University Hospital of Basel, Department of Thoracic Surgery, Basel, Switzerland